CLINICAL TRIAL: NCT07142083
Title: Comparison of the Effects of Bioelectrical Impedance Analysis-Guided Versus Conventional Fluid Resuscitation Strategies on 28-Day Mortality in Intensive Care Unit Patients After Major Surgery
Brief Title: BIA-Guided vs. Conventional Fluid Resuscitation in ICU Patients
Acronym: BIA-FLUID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Fatma ULGER, Ondokuz Mayıs University, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BIA2024
Record Dates: First submitted 2025-08-06; First posted 2025-08-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Fluid and Electrolyte Imbalance; Anesthesia
Keywords: Bioelectrical impedance analysis; Intensive Care; Fluid Resuscitation; Postoperative Fluid Management

STUDY DESIGN:
Intervention Model Description: A computer-generated block randomization list will be created using an online randomization tool by a researcher who is not involved in patient treatment or follow-up. Patients will be assigned to one of two groups (BIA-guided fluid management or conventional fluid therapy) based on sealed opaque envelopes prepared in advance according to the randomization sequence.
Who Masked: Investigator, Outcomes Assessor
Masking Description: To preserve the integrity of the study results, group assignments (BIA-guided fluid resuscitation vs. conventional fluid resuscitation) were concealed from the clinical staff involved in patient care and data collection. In addition, the investigators responsible for evaluating the primary and secondary outcomes (outcome assessors) were blinded to group allocation. Prior to participation, all patients or their legal representatives were thoroughly informed about the study's purpose, the nature of the two fluid management strategies, the randomization process, and the blinding of group information. Informed consent was obtained after ensuring full understanding of the methodology, including the confidentiality of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIA-Guided Fluid Therapy (Experimental): Patients in this group will receive postoperative fluid therapy guided by bioelectrical impedance analysis (BIA) using the Body Composition Monitor (BCM) device. Daily fluid decisions will be based on measurements such as Extracellular water (ECW)/ Total body water (TBW) and phase angle.
  Interventions: Device: Bioelectrical Impedance Analysis (BCM)
- Conventional Fluid Therapy (Active Comparator): Patients in this group will receive conventional fluid management based on routine clinical parameters, including vital signs, urine output, physical examination, and laboratory values. No bioelectrical impedance analysis will be performed in this group.
  Interventions: Procedure: Conventional Fluid Management

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis (BCM) — The Body Composition Monitor (BCM) device will be used to perform daily bioelectrical impedance measurements to guide fluid resuscitation in critically ill patients after major surgery. Measurements include extracellular water, intracellular water, total body water, and phase angle. The results will be used to tailor fluid therapy.
  Arms: BIA-Guided Fluid Therapy
Procedure: Conventional Fluid Management — Patients in this group will receive fluid therapy based on standard clinical parameters including blood pressure, heart rate, urine output, laboratory values, and physical examination. No bioelectrical impedance measurement will be performed.
  Arms: Conventional Fluid Therapy

SUMMARY:
In this study aimed to compare bioelectrical impedance analysis (BIA)-guided fluid resuscitation with conventional fluid management strategies in patients admitted to the intensive care unit (ICU) following major surgery. The primary objective is to evaluate whether BIA-guided fluid therapy reduces 28-day mortality by optimizing fluid balance and preventing volume-related complications. Secondary outcomes include cumulative fluid balance, ICU and hospital length of stay, duration of mechanical ventilation, and need for vasopressor or inotropic support. This study is expected to provide evidence for the clinical utility and applicability of BIA in guiding postoperative fluid therapy in critically ill patients.

DETAILED DESCRIPTION:
Fluid resuscitation plays a critical role in the perioperative care of patients undergoing major surgery.

Traditionally, fluid therapy decisions in the intensive care unit (ICU) have relied on static clinical parameters, which may not always reflect the patient's actual volume status. Bioelectrical impedance analysis (BIA) offers a noninvasive and dynamic assessment of hydration status, enabling more precise fluid management tailored to individual needs. This prospective, randomized controlled study aims to compare BIA-guided fluid resuscitation with conventional fluid management strategies in postoperative ICU patients. A total of 80 adult patients who meet the inclusion criteria will be randomized into two groups. Group 1 will receive standard fluid therapy based on clinical evaluation, including heart rate, blood pressure, urine output, passive leg raising test, and vena cava ultrasound assessment. Group 2 will undergo BIA measurements at 0, 12, 24, and 48 hours post-ICU admission to guide fluid management according to hydration status (dehydrated, euvolemic, or hypervolemic). The primary outcome is 28-day all-cause mortality. Secondary outcomes include cumulative fluid balance, ICU and hospital length of stay, duration of mechanical ventilation, and need for vasopressors or inotropic agents. By evaluating clinical outcomes between the two approaches, this study seeks to determine whether BIA-guided fluid management offers a clinically meaningful advantage in postoperative critical care.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing major surgery under general anesthesia(Major surgery defined as: vascular clamping or organ ischemia, intraoperative blood loss >1000 mL, need for >10 mcg/min norepinephrine infusion, surgery duration >4 hours, or requirement for perioperative blood transfusion)
* Admission to the intensive care unit (CU) after surgery
* Informed consent obtained

Exclusion Criteria:

* Refusal to participate or failure to provide informed consent
* Undergoing laparoscopic or emergency surgery
* Severe major organ dysfunction:Acute kidney injury stage 2 or 3 (KDIGO 2012) • Acute or chronic liver failure (ALT >3x or Child A-C cirrhosis
* Conditions preventing accurate BIA measurement: • Limb amputation • Metallic cardiac or joint prostheses • Pacemakers or intracardiac stents
* Body mass index >35 kg/m or < 18 kg/m
* Contraindications to lactated Ringer's solution (e.g. hypercalcemia, increased intracranial pressure)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | postoperative 28 days
  The number of participants in each group who die from any cause within 28 days after admission to the intensive care unit (ICU) following major surgery. The primary comparison will be between patients receiving bioelectrical impedance analysis (BIA)-guided fluid therapy and those receiving conventional fluid management.

SECONDARY OUTCOMES:
Cumulative fluid balance | First 48 hours after ICU admission
  Total fluid input minus total fluid output calculated cumulatively for each patient during ICU stay. Fluid balance will be recorded daily and evaluated within the first 48 hours after ICU admission.
ICU length of stay | The time from admission to the ICU to the time of discharge to the hospital ward; during the hospital stay, an average of 28 days
  The number of days each patient remains in the intensive care unit after major surgery, from admission to discharge from the ICU.
Hospital length of stay | Measured in days admitted in the hospital, an average of 28 days
  The total number of days from the patient's admission to the hospital (including ICU and ward stay) until discharge or death.
Duration of mechanical ventilation | First 48 hours after ICU admission
  Total number of hours each patient remains on invasive mechanical ventilation during the first 48 hours of ICU follow-up.
Requirement for inotropic support | First 48 hours after ICU admission
  The number of patients in each group requiring any inotropic or vasopressor therapy during the ICU stay. The type, dose, and duration of inotropic support will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ülger, Study Director — Ondokuz Mayıs University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical restrictions and the absence of prior informed consent for data sharing. Additionally, the study does not include a data sharing provision in the approved protocol or institutional ethics approval.

REFERENCES:
- [Background] Chung YJ, Kim EY. Usefulness of bioelectrical impedance analysis and ECW ratio as a guidance for fluid management in critically ill patients after operation. Sci Rep. 2021 Jun 9;11(1):12168. doi: 10.1038/s41598-021-91819-7. PMID 34108597
- [Background] Myatchin I, Abraham P, Malbrain MLNG. Bio-electrical impedance analysis in critically ill patients: are we ready for prime time? J Clin Monit Comput. 2020 Jun;34(3):401-410. doi: 10.1007/s10877-019-00439-0. Epub 2019 Dec 5. No abstract available. PMID 31808061
- [Background] Wang K, Sun SL, Wang XY, Chu CN, Duan ZH, Yang C, Liu BC, Ding WW, Li WQ, Li JS. Bioelectrical impedance analysis-guided fluid management promotes primary fascial closure after open abdomen: a randomized controlled trial. Mil Med Res. 2021 Jun 7;8(1):36. doi: 10.1186/s40779-021-00329-0. PMID 34099065
- [Background] Basso F, Berdin G, Virzi GM, Mason G, Piccinni P, Day S, Cruz DN, Wjewodzka M, Giuliani A, Brendolan A, Ronco C. Fluid management in the intensive care unit: bioelectrical impedance vector analysis as a tool to assess hydration status and optimal fluid balance in critically ill patients. Blood Purif. 2013;36(3-4):192-9. doi: 10.1159/000356366. Epub 2013 Dec 20. PMID 24496190